CLINICAL TRIAL: NCT00472160
Title: Preoxygenation Using Noninvasive Ventilation Prior Intubation in Hypoxemic Patients
Brief Title: Preoxygenation Using NIV in Hypoxemic Patients
Acronym: PREOXY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Cecile JOURDAIN, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P060230
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2007-05

CONDITIONS: Critical Illness; Hypoxemia
Keywords: Preoxygenation; Non Invasive Ventilation; Continuous Positive Airway Pressure,; Intubation,; Organ failure
MeSH Terms: conditions — Critical Illness; Hypoxia | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Non Invasive Ventilation
  Interventions: Procedure: Non Invasive Ventilation

INTERVENTIONS:
Procedure: Non Invasive Ventilation — Non Invasive Ventilation

SUMMARY:
Critically ill patients are predisposed to oxyhaemoglobin desaturation during intubation. For the intubation of hypoxemic patients, preoxygenation using non invasive ventilation (NIV) is more effective at reducing arterial oxyhaemoglobin desaturation than standard method.

Objectives: To find out whether NIV, as a preoxygenation method, is more effective at reducing the degree of organ dysfunction/failure than standard preoxygenation during the week following endotracheal intubation.

DETAILED DESCRIPTION:
During the inclusion period (at least 10 min and maximum 30 min), the patients ware a high FiO2 mask, driven by 10-15L/min oxygen and are randomly assigned to control or NIV group. Preoxygenation is then performed for a 3 minute period prior to a standardized rapid sequence intubation. For the control group, preoxygenation use a non-re-breather bag-valve mask driven by 15L/min oxygen. Patients allow to breath spontaneously with occasional assists (usual preoxygenation method). For the NIV group, pressure support mode is delivered by an ICU ventilator through a face mask adjusted to obtain an expired tidal volume of 7 to 10 mL/kg. The fraction of inspired oxygen (FiO2) was 100% and we used a PEEP level of 5 cmH2O.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients with acute respiratory failure requiring intubation

Exclusion Criteria:

* Encephalopathy or coma, cardiac resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The maximum Sequential organ failure assessment (SOFA) score observed during the first week following endotracheal intubation. | the first week

SECONDARY OUTCOMES:
The mean drop in SpO2 during endotracheal intubation. | during the intubation
Number of organ failures (SOFA score >2) | during the 7 days after intubation
ICU length of stay | during the stay in reanimation
Mortality | in reanimation

CONTACTS AND LOCATIONS:
Overall Officials: Christophe BAILLARD, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital de Bobigny, Bobigny, France

REFERENCES:
- [Result] Baillard C, Fosse JP, Sebbane M, Chanques G, Vincent F, Courouble P, Cohen Y, Eledjam JJ, Adnet F, Jaber S. Noninvasive ventilation improves preoxygenation before intubation of hypoxic patients. Am J Respir Crit Care Med. 2006 Jul 15;174(2):171-7. doi: 10.1164/rccm.200509-1507OC. Epub 2006 Apr 20. PMID 16627862
- [Derived] Baillard C, Prat G, Jung B, Futier E, Lefrant JY, Vincent F, Hamdi A, Vicaut E, Jaber S. Effect of preoxygenation using non-invasive ventilation before intubation on subsequent organ failures in hypoxaemic patients: a randomised clinical trial. Br J Anaesth. 2018 Feb;120(2):361-367. doi: 10.1016/j.bja.2017.11.067. Epub 2017 Nov 23. PMID 29406184